CLINICAL TRIAL: NCT02969447
Title: Effect of Intra-venous Oxytocin Injection After Fetal Expulsion in Management of Third-stage of Labor After Second Trimester Medical Pregnancy Termination
Brief Title: Management of Third-stage of Labor After Second Trimester Medical Pregnancy Termination
Acronym: ANDDROID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2016/20
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Retained Placenta
Keywords: Retained Placenta; Second trimester medical termination; Third stage labor; Oxytocin
MeSH Terms: conditions — Placenta, Retained

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin administration after fetal expulsion (Experimental): Administration of 10 units of intra venous oxytocin after fetal expulsion
  Interventions: Drug: Administration of 10 units of intra venous oxytocin after fetal expulsion
- No additional medication after fetal expulsion (No Intervention)

INTERVENTIONS:
Drug: Administration of 10 units of intra venous oxytocin after fetal expulsion
  Arms: Oxytocin administration after fetal expulsion

SUMMARY:
Prospective randomized trail which compare 2 regimens for third-stage management after second trimester medical pregnancy termination : 10UI intra venous oxytocin or no additional medication after fetal expulsion. Primary outcome was the incidence of placental retention.

DETAILED DESCRIPTION:
Complication of third stage of labor in second trimester medical pregnancy termination is not well studied. Accord to publications, the placental retention rate is 30 to 40% in these situations. Placental retention may be associated with increased blood loss, increased requirement for blood transfusion anesthetic and operative complications, and infectious morbidity. The high incidence of retained placenta is an area of clinical concern. Publications reveal a wide variation in practices but there are only few studies about third stage of labor in second trimester medical pregnancy termination. The study is a prospective randomized trial. Two third stage management strategies are compared: 10 units of intra venous oxytocin (group 1) and no additional medication (group 2) after fetal expulsion. It concerns pregnancies between 14 and 28 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* medical pregnancy termination between 14 and 28 weeks gestation
* informed consent obtained

Exclusion Criteria:

* less than 18 years old
* refusal to consent
* in utero fetal death

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Incidence of placental retention | Up to 30 minutes after fetal expulsion

SECONDARY OUTCOMES:
Incidence of partial placental retention | Up to 1 hour after fetal expulsion
Incidence of digital exploration | Up to 1 hour after fetal expulsion
Incidence of blunt curettage | Up to 1 hour after fetal expulsion
Incidence of post-partum hemorrhage | Up to 1 hour after fetal expulsion
Blood loss | Up to 1 hour after fetal expulsion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided